CLINICAL TRIAL: NCT00192439
Title: A Study to Describe the Incidence Rate and Clinical Features of Human Meta Pneumovirus (hMPV) Infection of the Lower Respiratory Tract in Hospitalized Children at High Risk for Severe Disease
Brief Title: Study to Evaluate the Human Infection of the Lower Respiratory Tract in Children at High Risk
Status: Completed | Type: Observational
Sponsor: MedImmune LLC (Industry)
Other Study IDs: MI-CP096
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Severe Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Behavioral: High Risk Respiratory Disease

SUMMARY:
- Estimate the incidence rate of hMPV infection detected by RT-PCR from frozen nasal wash aspirates in children at high risk for severe LRI disease (hospitalized at <2 years of age).

DETAILED DESCRIPTION:
* A prospective, epdemiological study to estimate the incidence rate of hMPV infection as determined by RT-PCR from frozen nasal wash aspirates taken from children hospitalized with LRI who are at high risk for severe disease.
* No study drug will be administered for this study.

ELIGIBILITY:
Inclusion Criteria:

* Be premature (less than 36 weeks gestation) and less than or equal to 12 months of age, and/or
* Be less than or equal to 24 months of age with CHD (other than uncomplicated small atrial or ventricular septal defects or patent ductus arteriosus) that is judged to be hemodynamically significant, and/or
* Be less than or equal to 24 months of age with CLD of prematurity (BPD) requiring medical intervention/management (i.e., supplemental oxygen, steroids, bronchodilators, or diuretics within the previous 6 months).
* Hospital admission diagnosis referable to an acute lower respiratory tract infection or cardio/respiratory illness with a presumed respiratory infection (e.g., bronchiolitis, bronchitis, or pneumonia or cardiac decompensation associated with respiratory infection); admission must occur between October 1 and June 30 for northern hemisphere sites, and between March 1 and November 30 for southern hemisphere sites.
* Study enrollment within 2 days after hospitalization.
* Admission from the community to the Pediatric ward, Neonatal Intensive Care Unit, or the Intensive Care Unit.
* Have written informed consent obtained from the parent or legal guardian prior to study entry.

Exclusion Criteria:

* Known HIV infection or a mother with known HIV infection.

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1500 (Actual)
Dates: Start 2003-12; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Gomez, M.D., Study Director — MedImmune LLC
Locations (24):
- United States (16):
  - Miller Children's Hospital, Long Beach, California
  - The Children's Hospital, Denver, Colorado
  - Children's Memorial Hospital, Chicago, Illinois
  - New England Medical Center, Boston, Massachusetts
  - The Children's Hospital, Buffalo, New York
  - Schneider Children's Hospital, Long Island Jewish Medical Center, New Hyde Park, New York
  - Univ. of Rochester Medical Center, Rochester, New York
  - Suny Upstate Medical Univ., Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Univ. School of Medicine, Winston-Salem, North Carolina
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Dept. of Pediatrics, Providence, Rhode Island
  - Lebonheur Children's Medical Center, Memphis, Tennessee
  - Univ. of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Children's Hospital and Regional Medical Center, Seattle, Washington
- Australia (3):
  - University Dept. of Paediatrics, Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Murdoch Children's Research Institute, Parkville, Victoria
  - University of Western Australia, Perth, Western Australia
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - Univ. of Mannitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - The Hospital for Sick Children, Toronto, Ontario
- Institute of Pediatrics, University of Milan, Milan, Italy